CLINICAL TRIAL: NCT04710108
Title: Testing Message Modality of Culturally Appropriate Nutrition Communication for Mexican American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Merced (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A. Susana Ramirez, Associate Professor, University of California, Merced
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K01CA190659-5; K01CA190659 (NIH)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Sugar Sweetened Beverage Consumption; Nutrition; Lifestyle-related Condition; Lifestyle Risk Reduction
Keywords: Values-based messages; Message modality; Health communication
MeSH Terms: conditions — Mental Disorders; Risk Reduction Behavior | interventions — Health Communication

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No treatment control (No Intervention): No treatment; no intervention (survey only)
- Video (Experimental): A Taste of Home video, Poet: Monica Mendoza (spoken word poem from The Bigger Picture; images of Hispanic female poet interspersed with images of environment)
  Interventions: Other: Health Communication
- Print (Experimental): A Taste of Home comic book, Poet: Monica Mendoza (spoken word poem from The Bigger Picture; images of Hispanic female poet interspersed with images of environment)
  Interventions: Other: Health Communication

INTERVENTIONS:
Other: Health Communication — Spoken word poem set to video images performed by author. Comic book was transformed from the video that was equivalent in content to the video.
  Other Names: Values based messaging about sugar sweetened beverages
  Arms: Print; Video

SUMMARY:
A randomized controlled trial to test the effects of culturally appropriate nutrition communication delivered via different modalities for Mexican American women.

DETAILED DESCRIPTION:
A randomized controlled trial with pre-test and immediate post-test was employed to test the effects of different types of message modalities (video vs. comic book). The study was conducted online with Mexican American women aged 18-29 years old. Messages focused on sugary beverage consumption and the main outcomes are individual intention to adopt health behaviors which will be measured by the increased degree of individual knowledge, attitudes, subjective norms, self-efficacy, and intention to reduce SSB consumption, as well as social level behavior changes that will be measured by the improved magnitude of public health literacy, SSB media literacy, and empowerment. Secondary outcomes of interest include the evaluations on the dimension of message themselves include participants' direct reaction to messages and their perceived effectiveness of messages, which will be measured by transportation of messages, identification of characters, emotional response of scenes, perceived effectiveness of messages, engagement with messages, and willingness to disseminate messages.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Latina or Hispanic
* Self-identify as a woman
* Self-reported as being of age between 18-29 years

Exclusion Criteria:

* Not Mexican American (defined as having at least 1 grandparent born in Mexico or self-identifying as Mexican or Mexican American)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as women
Enrollment: 129 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Knowledge | Immediately post-intervention exposure
  Knowledge increases self-efficacy and makes people to make better health choices for themselves and knowledge of the negative consequences of a given health behavior increases the intention to reduce that behavior. Therefore, better knowledge of the negative consequences of SSB consumption directly impacts individual level SSB consumption. We created an SSB knowledge scale comprising 6 true or false items adapted from multiple studies. The statements are as follows: "Excessive sugar consumption causes (1) health problems (2) weight gain (3) dental caries (4) diabetes (5) cancer and (6) heart disease." Greater scores on this scale represented greater levels of SSB knowledge.
Attitude toward sugary beverage consumption | Immediately post-intervention exposure
  The theory of planned behavior (TPB) states that attitude toward reducing SSB consumption is an individual level outcome predicting intention to reduce SSB consumption. We will measure attitude toward reducing SSB consumption as a single, 5-point Likert item with responses ranging from Very Good=5 to Very Bad=1 as follows: "Reducing my consumption of sugary beverages over the next 3 months would be." Greater scores on this scale represented more positive attitude toward reducing SSB consumption
Subjective norms toward sugary beverage consumption | Immediately post-intervention exposure
  The TPB states that subjective norms to reduce SSB consumption is an individual level outcome facilitating intention to reduce SSB consumption. We will measure intention to reduce SSB consumption as a single, 5-point Likert item with responses ranging from Strongly Agree=5 to Strongly Disagree=1 as follows: "Most people who are important to me would approve of my drinking less than 1 cup of sugary drinks each day for the next 3 months." Greater scores on this scale represented greater levels of intention to reduce SSB consumption.
Self-efficacy toward SSB consumption | Immediately post-intervention exposure
  The TPB states that self-efficacy to reduce SSB consumption is an individual level outcome predicting intention to reduce SSB consumption. We will measure self-efficacy to reduce SSB consumption as a single, 5-point Likert item with responses ranging from Strongly Agree=5 to Strongly Disagree=1 as follows: "If I really wanted to, I am confident that I could reduce my consumption of sugary beverages over the next 3 months." Greater scores on this scale represented greater levels of self-efficacy to reduce SSB consumption.
Intention to reduce SSB consumption | Immediately post-intervention exposure
  The TPB states that intention to reduce SSB consumption is an individual level outcome predicting actual reduction of SSB consumption. We will measure intention to reduce SSB consumption as a single, 5-point Likert item with responses ranging from Strongly Agree=5 to Strongly Disagree=1 as follows: "I plan to reduce my consumption of sugary beverages over the next 3 months." Greater scores on this scale represented greater levels of intention to reduce SSB consumption.
Media literacy | Immediately post-intervention exposure
  We will measure SSB related media literacy using a 5-point, 8-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1 adapted from Chen et. al.(Cronbach's Alpha = 0.83). This scale measures how much the participants understand the ways in which SSB industry used media to influence and manipulate their SSB consumption behaviors. Some sample items are as follows: "Certain sugary drink brands are designed to appeal to people like me," "Sugary drink ads show a healthy lifestyle to make people forget about the health risks, such as weight gain and diabetes" and "Sugary drink ads link drinking these beverages to things people want, like love, good looks, and power." Greater scores on this scale represent greater levels of SSB media literacy.
Public health literacy | Immediately post-intervention exposure
  Public health literacy is defined here as an understanding of the social determinants of health. We will measure it using a 5-point and 7-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1 (Cronbach's Alpha = 0.78). The seven items measure opinions about how much different external factors affect health because this best reflected an understanding of the social determinants of health: (1) money, (2) education, (3) safe and affordable housing, (4) early childhood experiences, and (5) government policies and programs (6) lifestyle choices and (7) consequences of system failure on the under-resourced. Greater scores on this scale represented greater levels of public health literacy.
Empowerment | Immediately post-intervention exposure
  Empowerment is defined as a social level construct measured using a 4-point and 8 item Likert scale adapted from Zimmerman et. al. with responses ranging from Strongly Agree/Very Effective=4 to Strongly Disagree/Not Effective at all=1. The scale comprised three subscales namely (1) Community control (2 items; Cronbach's Alpha = 0.68); (2) Perceived effectiveness of actions to influence community decisions (3 items; Cronbach's Alpha = 0.79); and (3) Perceived difficulty (3 items, Cronbach's Alpha = 0.78). Sample questions from each subscale were as follows: "I can influence decisions that affect my community," "How effective would it be to attend meetings about some community issue or problem in convincing public officials and institutions to do something?" and "Community problems are often so complicated that even informed people can't figure out what should be done about them." Greater scores on this scale represented greater levels of psychological empowerment.

SECONDARY OUTCOMES:
Transportation | Immediately post-intervention exposure
  We will measure transportation of messages using a 5-point, 2-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1 adapted based on scales by Green & Brock and Kim (Cronbach's Alpha = 0.85). The two items in the scale are, "I could picture myself in the scene of the events shown in the message," and "My attention was fully captured while viewing the message." Greater scores on this scale represent greater levels of engagement with the video.
Identification | Immediately post-intervention exposure
  Identification is measured using a 5-point, 4-item Likert scale adapted from scales by Cohen and Phua (Cronbach's Alpha = 0.84). Greater scores on this scale represent greater degree of identification with the character in the video. Identification with characters also include the perceived similarity with main character in the video, which will be measured using a 5-point, 2-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1 adapted from Cohen et. al. (Cronbach's Alpha = 0.93). The two items in the scale are, "I feel the person in the message, and I have many things in common," and "The person in the video and I are similar in many ways." Greater scores represent greater levels of perceived similarity.
Emotional response to video | Immediately post-intervention exposure
  We will measure emotional responses to the video using a 11-item, 5-point scale with responses ranging from Not at all=1 to Extremely=5 adapted from Dixon et. al. (Cronbach's Alpha = 0.95). The question stated "We are interested in how this message made you feel. Please indicate the extent to which the message made you feel…" The scale consisted of seven negative emotions viz., Disgusted, Anxious, Ashamed, Fearful, Guilty, Sad and Angry and four positive emotions viz., Proud, Validated, Hopeful and Empathetic. Higher scores on this scale represented more positive emotional response to the video.
Perceived effectiveness | Immediately post-intervention exposure
  Perceived effectiveness of the message is known to affect intention to engage in a given health behavior. Furthermore, some researchers have raised concerns of reactance as a negative consequence of persuasive messages69, 70 while others seem to argue that it does not necessarily affect the efficacy of a message. Therefore, we will measure perceived effectiveness of and reactance to the stimuli as a proxy measure for intention to reduce SSB consumption using a 5-point, 14-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1 adapted from Dixon et. al and other prior research. This scale comprised 4 subscales namely (1) Message Acceptance (2 items, Cronbach's Alpha = 0.89); (2) Argument Strength (4 items, Cronbach's Alpha = 0.88); (3) Personalized Perceived Effectiveness (7 items, Cronbach's Alpha = 0.91); and (4) Reactance (1 item). Greater scores on this scale represented greater levels of perceived effectiveness of the message.
Willingness to disseminate the message | Immediately post-intervention exposure
  We will measure the willingness to disseminate the message by a 10-point Net Promoter Score (NPS) adapted from Alismail et. al (Cronbach's Alpha = 0.87). The item is, "On a scale from 0-10, how likely are you to recommend this message to a friend or family". Greater scores on this scale indicate greater willingness to recommend the message to others.
Engagement with the message | Immediately post-intervention exposure
  Engagement with message in this study means engagement with The Bigger Picture Project campaign since the two experimental treatments were all from this campaign. We will measure this outcome by clicking the campaign link for more information in Qualtrics shown on the stimuli display pages with clicked = 1 and did not click = 0.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Ramirez, Principal Investigator — University of California, Merced
Locations (1):
- University of California Merced SONA System (Online Platform), Merced, California, United States

IPD SHARING:
Plan to Share IPD: No